CLINICAL TRIAL: NCT00406237
Title: Open Label, Single Dose Study Of The Pharmacokinetics Of Tigecycline In Adult Subjects With Primary Biliary Cirrhosis
Brief Title: Pharmacokinetic Study Of Tigecycline In Adult Subjects With Primary Biliary Cirrhosis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: 3074A1-120; B1811005
Record Dates: First submitted 2006-11-29; First posted 2006-12-04 (Estimated); Last update posted 2011-04-04 (Estimated); Status verified 2011-04

CONDITIONS: Liver Cirrhosis, Biliary
MeSH Terms: conditions — Liver Cirrhosis, Biliary | interventions — Tigecycline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: tigecycline

INTERVENTIONS:
Drug: tigecycline — Single intravenous dose of tigecycline 50 mg, as a 30-minute infusion
  Other Names: Tygacil, GAR-936

SUMMARY:
Open label, single dose study of the pharmacokinetics of tigecycline in adult subjects with primary biliary cirrhosis (PBC)

DETAILED DESCRIPTION:
pharmacokinetic study

ELIGIBILITY:
Inclusion Criteria:

* Men and nonlactating and nonpregnant women greater than or equal to 18 years of age
* Subjects with biopsy proven primary biliary cirrhosis (PBC) disease in the asymptomatic or symptomatic phase of PBC.
* Otherwise healthy as determined by the investigator on the basis of medical history, physical examination, clinical laboratory test results (other than those associated with PBC), vital signs, and 12-lead electrocardiogram (ECG).

Exclusion Criteria:

* Subjects with a recent increase in bilirubin, bilirubin >15 mg/dL, presence of ascites, esophageal varices, or hepatic encephalopathy.
* Any major illness that in the investigator's judgment will substantially increase the risk associated with the subject's participation in the study
* Any malignancy including hepatocellular carcinoma.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2006-12; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
To assess the pharmacokinetics (PK) of tigecycline in subjects with cholestatic hepatic dysfunction. | 5 days

SECONDARY OUTCOMES:
To assess the safety and tolerability of single doses of tigecycline in subjects with cholestatic hepatic dysfunction. | 15 days

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (3):
- United States (2):
  - Pfizer Investigational Site, Saint Paul, Minnesota
  - Pfizer Investigational Site, Durham, North Carolina
- Pfizer Investigational Site, Santurce, Puerto Rico, Puerto Rico

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=3074A1-120&StudyName=Pharmacokinetic%20Study%20Of%20Tigecycline%20In%20Adult%20Subjects%20With%20Primary%20Biliary%20Cirrhosis